CLINICAL TRIAL: NCT06422052
Title: Epidemiological Investigation of Helicobacter Pylori-infected Patients and the Effect of Eradication Treatment on Dyspepsia Symptoms
Status: Recruiting | Type: Observational
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Hong Lu, MD, Medical Doctor of Division of Gastroenterology and Hepatology of Renji Hospital,Professor of Medicine, RenJi Hospital
Other Study IDs: rjhy20240504
Record Dates: First submitted 2024-05-14; First posted 2024-05-20 (Actual); Last update posted 2024-12-30 (Actual); Status verified 2024-11

CONDITIONS: Helicobacter Pylori Infection; Dyspepsia
Keywords: Helicobacter Pylori Infection; Dyspepsia
MeSH Terms: conditions — Dyspepsia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Dyspepsia with Helicobacter pylori infection
  Interventions: Other: Epidemiological questionnaire and Functional Dyspepsia Symptom Diary（FDSD）

INTERVENTIONS:
Other: Epidemiological questionnaire and Functional Dyspepsia Symptom Diary（FDSD） — H. pylori infection was confirmed by 13C/ 14C-breath test and/or rapid urease test under endoscopy and histopathological examination. Epidemiological questionnaire and Functional Dyspepsia Symptom Diary (FDSD) were used to investigate basic information and assess dyspeptic symptoms. Patients with dyspepsia who successfully eradicated Helicobacter pylori infection will be followed up for dyspeptic symptoms after 2 months and 6 months to evaluate the relief of dyspeptic symptoms.

SUMMARY:
The objectives of this multicenter, prospective, observational study were to investigate the incidence of dyspeptic symptoms in patients with Helicobacter pylori (H. pylori) infection and to continuously follow up the remission of dyspeptic symptoms after H. pylori eradication, so as to provide reference for the clinical diagnosis and treatment strategies of patients with H. pylori infection and dyspeptic symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged 18-80 years
* H. pylori infection diagnosed by 13C/ 14C-UBT (> 2 times the cutoff value) and/or gastroscopy (rapid urease strong positive and histological positive)
* Treatment-naive patients with Helicobacter pylori
* Ability and willingness to participate in the study and to sign and give informed consent

Exclusion Criteria:

* Under 18 or over 80 years old
* Organic digestive diseases, such as active peptic ulcer, gastroesophageal reflux, gastrointestinal bleeding, acute/chronic pancreatitis, acute/chronic cholecystitis, gallstones, intestinal obstruction, inflammatory bowel disease, etc.
* Combined with melena, hematemesis, anemia, emaciation and other alarm symptoms
* Pregnant and lactating women
* History of cancer
* History of subtotal gastrectomy
* Severe organ dysfunction of heart, liver, kidney, lung and other important organs and congenital diseases, such as grade IV heart failure, liver failure, uremia, respiratory failure, hemophilia, Wilson's disease, etc.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population targets male and female patients aged 15-80 who have not previously been treated for Helicobacter pylori and have been diagnosed via 13C/14C urea breath test or gastroscopy. Participants must be willing and able to give informed consent. Exclusions include individuals under 18 or over 80, those with organic digestive diseases, pregnant or nursing women, those with a history of cancer or partial gastrectomy, and individuals with severe organ dysfunction or congenital diseases. Also excluded are those with symptoms like melena, hematemesis, anemia, or cachexia.
Sampling Method: Non-Probability Sample
Enrollment: 2242 (Estimated)
Dates: Start 2024-03-11 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
the incidence of dyspepsia in patients with Helicobacter pylori infection | Time 0 when finished the Epidemiological questionnaire and Functional Dyspepsia Symptom Diary
  Proportion of patients with Helicobacter pylori infection with dyspeptic symptoms
Relief of Helicobacter pylori related dyspepsia | Patients with dyspepsia who have successfully eradicated Helicobacter pylori infection will be followed up for dyspepsia symptoms after 2 months and after 6 months to assess the remission of dyspepsia symptoms
  The Functional Dyspepsia Symptom Diary (FDSD) will be used to evaluate the dyspepsia symptoms of the patients

CONTACTS AND LOCATIONS:
Locations (26):
- China (26):
  - Chongqing Daping Hospital, Chongqing, Chongqing Municipality
  - The Ninth People's Hospital of Chongqing, Chongqing, Chongqing Municipality
  - The People's Hospital of Kaizhou District, CQ, Chongqing, Chongqing Municipality
  - The First Affiliated Hospital of Xiamen University, Xiamen, Fujian
  - The People's Hospital of Wuwei, Wuwei, Gansu
  - The First People's Hospital of Qinzhou, Qinzhou, Guangxi
  - The First Affiliated Hospital of Henan University of Science and Technology, Luoyang, Henan
  - Yongcheng People's Hospital of Henan Province, Shangqiu, Henan
  - Xuchang Central Hospital, Xuchang, Henan
  - Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Baotou Central Hospital, Baotou, Inner Mongolia
  - Dalian Friendship Hospital, Dalian, Liaoning
  - The First Affiliated Hospital of Dalian Medical University, Dalian, Liaoning
  - Renji Hospital, School of Medicine, Shanghai Jiao Tong University, Shanghai, Shanghai Municipality
  - Ruijin Hospital Luwan Branch, Shanghai, Shanghai Municipality
  - Shanghai Construction Group Hospital, Shanghai, Shanghai Municipality
  - Shanghai East Hospital, Shanghai, Shanghai Municipality
  - Shanghai Putuo Liqun Hospital, Shanghai, Shanghai Municipality
  - Shanghai Songjiang Central Hospital, Shanghai, Shanghai Municipality
  - West China Fourth Hospital, Sichuan University, Chengdu, Sichuan
  - First Teaching Hospital of Tianjin University of Traditional Chinese Medicine, Tianjing, Tianjing
  - The Second People's Hospital of Kashgar, Xinjiang, Kashgar, Xinjiang
  - Second People's Hospital of Jinning District, Kunming City, Kunming, Yunnan
  - Ningbo Hangzhou Bay Hospital, Ningbo, Zhejiang
  - The People's Hospital of Shengzhou, Ningbo, Zhejiang
  - Shengzhou People's Hospital, Shaoxing, Zhejiang

IPD SHARING:
Plan to Share IPD: No